CLINICAL TRIAL: NCT00380237
Title: Phase 1 Inpatient Study of the Safety and Immunogenicity of H9N2 (6-2) AA ca Reassortant (A/Chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca), a Live Attenuated Virus Vaccine Candidate for Prevention of Avian Influenza H9N2 Infection in the Event of a Pandemic (Study B)
Brief Title: Safety of and Immune Response to a Bird Flu Virus Vaccine (H9N2) in Healthy Adults (Study B)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Ruth Karron, MD, Center for Immunization Research, Johns Hopkins Bloomberg School of Public Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIR 211 (Study B); CHR H.22.05.03.11.B2
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Last update posted 2008-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Influenza; Virus Diseases
Keywords: Bird Flu; Avian Flu
MeSH Terms: conditions — Influenza, Human; Virus Diseases; Influenza in Birds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Two vaccinations with H9N2 (6-2) AA ca Reassortant (A/chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca) vaccine at a dose of 10^7 TCID50 delivered by nose drops. The second vaccination will be given 4 to 12 weeks after the first.
  Interventions: Biological: H9N2 (6-2) AA ca Reassortant (A/Chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca)

INTERVENTIONS:
Biological: H9N2 (6-2) AA ca Reassortant (A/Chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca) — Live attenuated H9N2 (6-2) AA ca Reassortant (A/Chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca) vaccine

SUMMARY:
Avian influenza (AI), also known as bird flu, has become a major public health concern in many regions of the world. The purpose of this study is to evaluate the safety of and immune response to an AI vaccine in healthy adults.

DETAILED DESCRIPTION:
AI is caused by a virus that occurs naturally among birds. Because the virus has the ability to mutate into a form that can efficiently spread among the human population, AI has the potential to cause pandemics. The purpose of this study is to evaluate the safety of and immune response to the AI vaccine H9N2 (6-2) AA ca Reassortant (A/Chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca) in healthy adults who have never been exposed to the H9N2 virus.

This study will last from approximately 6 weeks, up to a maximum of approximately 20 weeks. Participation includes a 10-day minimum hospital stay in an isolation unit of the Bayview Medical Center of Johns Hopkins University. Participants will be admitted to the isolation unit 2 days prior to vaccination. At vaccination, participants will be given one dose of the H9N2 (6-2) AA ca Reassortant (A/Chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca) vaccine in the form of nose drops. Each day for the next 7 days, participants' vital signs will be monitored and nasal washes will be collected to test for the presence of vaccine virus. Participants may be discharged from the hospital after 3 consecutive negative viral cultures, but not before Day 7 after vaccination. Follow-up visits will occur on Days 21, 28, and 42, and will include blood collection and a physical exam.

Participants who received the first dose of the (A/Chicken/Hong Kong/G9/97 x A/Ann Arbor/6/60 ca) vaccine will be asked to receive a second dose of the vaccine 4 to 12 weeks after receiving the initial dose. Study procedures will be identical to those related to the first vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Born after 1968
* Good general health
* Available for the duration of the study
* Female participants must agree to use acceptable forms of contraception

Exclusion Criteria:

* Significant medical illness, physical examination findings, or urine or blood abnormalities
* Clinically significant neurologic, heart, lung, liver, rheumatologic, autoimmune, or kidney disease
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, may interfere with the study
* Previously enrolled in an H9N2 influenza vaccine study or in any other study of a bird flu vaccine
* Positive for the H9N2 influenza A virus (serum hemagglutination inhibiting [HI] factor antibody titer greater than 1:8)
* Medical, work, or family problems as a result of alcohol or illegal drug use within 12 months prior to study entry
* History of severe allergic reaction or anaphylaxis
* Current asthma or reactive airway disease within 2 years prior to study entry
* History of Guillain-Barre syndrome
* HIV-1 serotype positive
* Hepatitis C virus (HCV) positive
* Hepatitis B surface antigen positive
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs within 30 days prior to study entry. Participants who have used topical corticosteroids are not excluded.
* Live vaccine within 4 weeks prior to study entry
* Killed vaccine within 2 weeks prior to study entry
* Absence of spleen
* Blood products within 6 months prior to study entry
* Current smoker unwilling to stop smoking for the duration of the study
* Plans to travel to the Southern Hemisphere or Asia within 14 days prior to study entry
* Plans to travel on a cruise ship within 14 days prior to study entry
* Work in the poultry industry
* Received an investigational agent within 30 days prior to study entry
* Allergy to eggs or egg products
* Purified protein derivative (PPD) positive (positive tuberculosis [TB] test)
* Family member with immunodeficiency
* Other condition that, in the opinion of the investigator, would affect participation in the study
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Safety, as defined by frequency of vaccine-related reactogenicity events and other adverse events (AEs) for each dose | Throughout study
Immunogenicity, as determined by antibody to H9N2 | At Days 0, 28, and 42
Determining the amount of serum and nasal wash antibody induced by the vaccine | Throughout study

SECONDARY OUTCOMES:
To determine the number of vaccinees infected with the H9N2 G9/AA ca reassortant vaccine candidate | Throughout study
To determine the phenotypic stability of vaccine virus shed | Throughout study
To develop a serum bank so that the capacity of the H9N2 G9/AA ca reassortant vaccine candidate to elicit HI and neutralizing antibodies to future H9N2 influenza viruses can be tested | Throughout study
To evaluate T-cell mediated and innate immune responses against the H9N2 G9/AA ca reassortant vaccine candidate | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research Inpatient Unit, Mason F. Lord Building, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Choi YK, Ozaki H, Webby RJ, Webster RG, Peiris JS, Poon L, Butt C, Leung YH, Guan Y. Continuing evolution of H9N2 influenza viruses in Southeastern China. J Virol. 2004 Aug;78(16):8609-14. doi: 10.1128/JVI.78.16.8609-8614.2004. PMID 15280470
- [Background] Cox NJ, Subbarao K. Global epidemiology of influenza: past and present. Annu Rev Med. 2000;51:407-21. doi: 10.1146/annurev.med.51.1.407. PMID 10774473
- [Background] Li C, Yu K, Tian G, Yu D, Liu L, Jing B, Ping J, Chen H. Evolution of H9N2 influenza viruses from domestic poultry in Mainland China. Virology. 2005 Sep 15;340(1):70-83. doi: 10.1016/j.virol.2005.06.025. PMID 16026813
- [Background] Lin YP, Shaw M, Gregory V, Cameron K, Lim W, Klimov A, Subbarao K, Guan Y, Krauss S, Shortridge K, Webster R, Cox N, Hay A. Avian-to-human transmission of H9N2 subtype influenza A viruses: relationship between H9N2 and H5N1 human isolates. Proc Natl Acad Sci U S A. 2000 Aug 15;97(17):9654-8. doi: 10.1073/pnas.160270697. PMID 10920197